CLINICAL TRIAL: NCT00797446
Title: A Clinical Outcomes Protocol of Photon/Proton Beam Radiation Therapy for Oropharyngeal Cancers
Brief Title: Photon/Proton Radiation Therapy for Oropharyngeal Cancers
Acronym: OP01
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment, feasibility issues
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI 0601-OP01
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Oropharyngeal Cancers
Keywords: Oropharyngeal; cancer; proton; radiation; outcomes
MeSH Terms: conditions — Oropharyngeal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Photon/Proton Radiation Therapy: Data collection will be obtained from the patient's medical records including initial evaluation, pathology report, dosimetry information, radiotherapy completion records and follow-up.

SUMMARY:
The purpose of this study is to collect information from the questionnaire and medical records to see what effects proton radiation has on cancer and collect and analyze morbidity outcomes: incidence of xerostomia (dry mouth) and tumor control.

DETAILED DESCRIPTION:
This is an outcomes study and is designed to collect information from the questionnaire and medical records to see what effects proton radiation has on cancer and collect and analyze morbidity outcomes: incidence of xerostomia (dry mouth) and tumor control.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven squamous cell carcinoma of oropharynx (tonsillar pillars, tonsillar fossa, soft palate, base of tongue).
* Stage-grouping:

  * Stage I (T1N0)
  * Stage II (T2N0)
  * Favorable Stage III (T1N1/T2N1) and selected stage IV (T1-T2 early N2b)2 or less lymph node and 2 or less cm diameter lymph node
  * Unfavorable stage III and selected stage IV (any T, N2c/N3)
* Surgery of the primary tumor/lymph nodes is limited to incisional/excisional biopsies.
* Will receive treatment with proton radiation.

Exclusion Criteria:

* Evidence of distant metastasis.
* Previous irradiation for head and neck cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Radiation Oncology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Collect and analyze morbidity outcomes: incidence of xerostomia | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months

SECONDARY OUTCOMES:
Collect and analyze tumor control outcomes. | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Roi Dagan, MD, MS, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parsons JT, Mendenhall WM, Stringer SP, Amdur RJ, Hinerman RW, Villaret DB, Moore-Higgs GJ, Greene BD, Speer TW, Cassisi NJ, Million RR. Squamous cell carcinoma of the oropharynx: surgery, radiation therapy, or both. Cancer. 2002 Jun 1;94(11):2967-80. doi: 10.1002/cncr.10567. PMID 12115386
- [Background] Mendenhall WM, Amdur RJ, Stringer SP, Villaret DB, Cassisi NJ. Radiation therapy for squamous cell carcinoma of the tonsillar region: a preferred alternative to surgery? J Clin Oncol. 2000 Jun;18(11):2219-25. doi: 10.1200/JCO.2000.18.11.2219. PMID 10829041
- [Background] Ojiri H, Mendenhall WM, Stringer SP, Johnson PL, Mancuso AA. Post-RT CT results as a predictive model for the necessity of planned post-RT neck dissection in patients with cervical metastatic disease from squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2002 Feb 1;52(2):420-8. doi: 10.1016/s0360-3016(01)02603-7. PMID 11872288
- [Background] Mendenhall WM, Villaret DB, Amdur RJ, Hinerman RW, Mancuso AA. Planned neck dissection after definitive radiotherapy for squamous cell carcinoma of the head and neck. Head Neck. 2002 Nov;24(11):1012-8. doi: 10.1002/hed.10187. PMID 12410537
- [Background] Doweck I, Robbins KT, Mendenhall WM, Hinerman RW, Morris C, Amdur R. Neck level-specific nodal metastases in oropharyngeal cancer: is there a role for selective neck dissection after definitive radiation therapy? Head Neck. 2003 Nov;25(11):960-7. doi: 10.1002/hed.10315. PMID 14603457
- [Background] Lefebvre JL, Chevalier D, Luboinski B, Kirkpatrick A, Collette L, Sahmoud T. Larynx preservation in pyriform sinus cancer: preliminary results of a European Organization for Research and Treatment of Cancer phase III trial. EORTC Head and Neck Cancer Cooperative Group. J Natl Cancer Inst. 1996 Jul 3;88(13):890-9. doi: 10.1093/jnci/88.13.890. PMID 8656441
- [Background] Brizel DM, Albers ME, Fisher SR, Scher RL, Richtsmeier WJ, Hars V, George SL, Huang AT, Prosnitz LR. Hyperfractionated irradiation with or without concurrent chemotherapy for locally advanced head and neck cancer. N Engl J Med. 1998 Jun 18;338(25):1798-804. doi: 10.1056/NEJM199806183382503. PMID 9632446
- [Background] Pignon JP, Hill C. Meta-analyses of randomised clinical trials in oncology. Lancet Oncol. 2001 Aug;2(8):475-82. doi: 10.1016/S1470-2045(01)00453-3. PMID 11905723
- [Background] Denis F, Garaud P, Bardet E, Alfonsi M, Sire C, Germain T, Bergerot P, Rhein B, Tortochaux J, Calais G. Final results of the 94-01 French Head and Neck Oncology and Radiotherapy Group randomized trial comparing radiotherapy alone with concomitant radiochemotherapy in advanced-stage oropharynx carcinoma. J Clin Oncol. 2004 Jan 1;22(1):69-76. doi: 10.1200/JCO.2004.08.021. Epub 2003 Dec 2. PMID 14657228
- [Background] Mendenhall WM, Parsons JT, Million RR, Cassisi NJ, Devine JW, Greene BD. A favorable subset of AJCC stage IV squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 1984 Oct;10(10):1841-3. doi: 10.1016/0360-3016(84)90259-1. No abstract available. PMID 6490417
- [Background] Mendenhall WM, Amdur RJ, Stringer SP, Villaret DB, Cassisi NJ. Stratification of stage IV SCC of the oropharynx. Head Neck. 2000 Sep;22(6):626-8. doi: 10.1002/1097-0347(200009)22:63.0.co;2-9. No abstract available. PMID 10941166
- [Background] Mancuso AA, Mukherji SK, Schmalfuss I, Mendenhall W, Parsons J, Pameijer F, Hermans R, Kubilis P. Preradiotherapy computed tomography as a predictor of local control in supraglottic carcinoma. J Clin Oncol. 1999 Feb;17(2):631-7. doi: 10.1200/JCO.1999.17.2.631. PMID 10080608
- [Background] Mendenhall WM, Parsons JT, Mancuso AA, Pameijer FJ, Stringer SP, Cassisi NJ. Definitive radiotherapy for T3 squamous cell carcinoma of the glottic larynx. J Clin Oncol. 1997 Jun;15(6):2394-402. doi: 10.1200/JCO.1997.15.6.2394. PMID 9196155
- [Background] Cooper JS, Fu K, Marks J, Silverman S. Late effects of radiation therapy in the head and neck region. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1141-64. doi: 10.1016/0360-3016(94)00421-G. PMID 7713779
- [Background] Korsten MA, Rosman AS, Fishbein S, Shlein RD, Goldberg HE, Biener A. Chronic xerostomia increases esophageal acid exposure and is associated with esophageal injury. Am J Med. 1991 Jun;90(6):701-6. PMID 2042685
- [Background] Eisbruch A, Ten Haken RK, Kim HM, Marsh LH, Ship JA. Dose, volume, and function relationships in parotid salivary glands following conformal and intensity-modulated irradiation of head and neck cancer. Int J Radiat Oncol Biol Phys. 1999 Oct 1;45(3):577-87. doi: 10.1016/s0360-3016(99)00247-3. PMID 10524409
- [Background] Mendenhall WM, Parsons JT, Cassisi NJ, Million RR. Squamous cell carcinoma of the tonsillar area treated with radical irradiation. Radiother Oncol. 1987 Sep;10(1):23-30. doi: 10.1016/s0167-8140(87)80066-x. PMID 3671769
- [Background] Peters LJ, Ang KK. The Role of Altered Fractionation in Head and Neck Cancers. Semin Radiat Oncol. 1992 Jul;2(3):180-194. doi: 10.1053/SRAO00200180. No abstract available. PMID 10717034
- [Background] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Background] Slater JD, Yonemoto LT, Mantik DW, Bush DA, Preston W, Grove RI, Miller DW, Slater JM. Proton radiation for treatment of cancer of the oropharynx: early experience at Loma Linda University Medical Center using a concomitant boost technique. Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):494-500. doi: 10.1016/j.ijrobp.2004.09.064. PMID 15890592
- [Background] Eisbruch A, Kim HM, Terrell JE, Marsh LH, Dawson LA, Ship JA. Xerostomia and its predictors following parotid-sparing irradiation of head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Jul 1;50(3):695-704. doi: 10.1016/s0360-3016(01)01512-7. PMID 11395238
- [Background] Pacholke HD, Amdur RJ, Morris CG, Li JG, Dempsey JF, Hinerman RW, Mendenhall WM. Late xerostomia after intensity-modulated radiation therapy versus conventional radiotherapy. Am J Clin Oncol. 2005 Aug;28(4):351-8. doi: 10.1097/01.coc.0000158826.88179.75. PMID 16062076
- [Result] Mendenhall WM, Stringer SP, Amdur RJ, Hinerman RW, Moore-Higgs GJ, Cassisi NJ. Is radiation therapy a preferred alternative to surgery for squamous cell carcinoma of the base of tongue? J Clin Oncol. 2000 Jan;18(1):35-42. doi: 10.1200/JCO.2000.18.1.35. PMID 10623691